CLINICAL TRIAL: NCT00527891
Title: Evaluation of the Signa Excite 3.0 T MRI Excite for Detection and Characterization of Liver Lesions
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2003-1051
Record Dates: First submitted 2007-09-10; First posted 2007-09-11 (Estimated); Last update posted 2012-07-31 (Estimated); Status verified 2012-07

CONDITIONS: Liver Cancer
Keywords: Liver Cancer; Magnetic Resonance Imaging; Signa Excite 3.0T MRI Scan
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Signa Excite 3.0 T MRI Scan: Signa Excite 3.0 T MRI Scan
  Interventions: Procedure: Signa Excite 3.0 T MRI Scan

INTERVENTIONS:
Procedure: Signa Excite 3.0 T MRI Scan — Signa Excite 3.0 T MRI scan within a two week period from the date of receiving standard 1.5 T MR of the liver area.

SUMMARY:
Primary Objective:

1. To compare the efficacy of 1.5T vs. 3T T1 and T2-weighted MR images sequences for the detection and evaluation of liver lesions.

DETAILED DESCRIPTION:
Magnetic resonance imaging is taken with scanners at different magnetic field strength. The current practice at UTMDACC is to perform these exams at 1.5 Tesla. Tesla is the unit of strength of the magnetic field. This study will compare the images taken at the standard 1.5 Tesla (T) magnetic field with those at the newer 3.0T magnetic field.

You are already scheduled to receive a standard 1.5 T MR of the liver area as requested by your doctor. As part of this study, you will then be asked to return on a separate date to have a similar exam performed with the Signal 3.0T Excite MR scanner. You will return within a two week period from the date of your first MRI examination. The examination will be performed in a machine that looks similar to the 1.5T scanner. It will also take about the same amount of time as the examination at 1.5T.

The images taken by both scanners will be evaluated and compared. After you have had the second scan, your participation in this study will be over. If there are new findings identified with the new scan your doctor will be notified.

This is an investigational study. The 3.0T scan will be performed free of charge. A total of 20 patients will take part in this study All will be enrolled at UTMDACC.

This protocol is partially funded by a research grant from General Electric Medical Systems (GEMS).

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a liver lesion larger than 1cm detected by a prior imaging modality.
2. Patients have been scheduled and are eligible for an MRI of the abdomen or MRI of the liver or MRI of the kidney examination.

Exclusion Criteria:

1) Patients who are unable to cooperate with breath hold.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients scheduled and are eligible for an MRI of the abdomen or MRI of the liver or MRI of the kidney examination at UT MD Anderson Cancer Center.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2004-06; Primary Completion 2007-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janio Szklaruk, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- U.T.M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center Website — http://www.mdanderson.org